CLINICAL TRIAL: NCT01018745
Title: Phase 1 Multiple Ascending Dose Study of BMS-907351 (XL184) Monotherapy in Japanese Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Multiple Ascending Dose Study of BMS-907351 (XL184) in Patients With Solid Tumors in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA205-001
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-907351 (XL184) (Experimental)
  Interventions: Drug: BMS-907351 (XL184)

INTERVENTIONS:
Drug: BMS-907351 (XL184) — Capsules, Oral, 25, 50, 75, 100, 125 and 175 mg, Once daily, Until disease progression or unacceptable toxicity became apparent

SUMMARY:
The purpose of this clinical study is to establish the maximum tolerated dose (MTD) and recommended Phase 2 dose (or dose range as appropriate) of BMS-907351 (XL184) when administered orally on a once daily schedule in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group performance 0-2

Exclusion Criteria:

* Subject has uncontrolled intercurrent illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To establish the MTD and recommended Phase 2 dose (or dose range as appropriate) of BMS-907351 (XL184) when administered orally on a once daily schedule in subjects with advanced or metastatic solid tumors | Within the first 28 days

SECONDARY OUTCOMES:
To assess the safety and tolerability of multiple doses of BMS-907351 (XL184) administered orally on a once daily schedule in subjects with advanced or metastatic solid tumors | Day 1, 2, 5, 8, 15, 19, 20, 29 and every 2 weeks thereafter
To assess plasma pharmacokinetics (PK) of oral administration of BMS-907351 (XL184) and the metabolite(s) in subjects with advanced or metastatic solid tumors | Day 1, 5, 15, 19 and 29
To assess tumor response (preliminary anti-tumor activity) after repeated administration of BMS-907351 (XL184) | Every 8 weeks
To assess the pharmacodynamic correlates of BMS-907351 (XL184) activity | Day 1, 5, 15, 19, 29 and every 4 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-Ku, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx